CLINICAL TRIAL: NCT00873197
Title: A Study to Assess the Pharmacokinetics, Tolerability and Safety of the Co-administration of Sancuso® (Transdermal Granisetron) and Intravenous Granisetron in Healthy Subjects
Brief Title: PK, Tolerability and Safety of the Co-administration of Sancuso® (Transdermal Granisetron) and IV Granisetron
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 392MD/41/C
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Co-administration of transdermal and intravenous granisetron; Granisetron; Healthy subjects; Intravenous; Pharmacokinetic profile; Sancuso® patch; Transdermal; Pharmacokinetics
MeSH Terms: interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sancuso® patch/IV granisetron (Experimental): Subjects will receive 1 Sancuso® patch worn for 7 days (168 hours). Immediately after the patch has been applied on Day 1, IV granisetron will be administered over 30 seconds. Following patch removal at 168 hours, a new patch will be immediately applied to the opposite arm and will remain in place for a further 7 days (168 to 336 hours).
  Interventions: Drug: granisetron

INTERVENTIONS:
Drug: granisetron — Sancuso® 3.1 mg/24 hours; transdermal. One patch applied to healthy intact skin on the upper outer arm and worn for 7 days (168 hours) followed by a second patch applied to the opposite arm at 168 hours for a further 7 days (168 to 336 hours).
  Kytril® (granisetron hydrochloride) 1 mg/mL; IV; 0.01 mg/kg (maximum 1 mg) administered over 30 seconds immediately following patch application on Day 1 only.
  Other Names: Granisetron Transdermal System; Sancuso® patch; Kytril®; Granisetron Injection

SUMMARY:
This study has been designed to investigate the pharmacokinetic and safety profile of the co-administration of intravenous (IV) and transdermal granisetron, as well as characterise the pharmacokinetics of multiple transdermal dosing.

DETAILED DESCRIPTION:
Sancuso® is designed to provide antiemetic prophylaxis for chemotherapy of up to 5 days duration. In exceptional clinical situations in which the patch is not applied at the appropriate time (i.e. 24-48 hours pre-chemotherapy), clinicians might use a single IV dose of granisetron to provide prophylaxis while the granisetron from the patch reaches a therapeutic plasma concentration.

Most chemotherapeutics are dosed in a single day, with a 2- or 3-week interval between doses; however, several regimens are administered over more than 5 days and others are given at frequencies (e.g. every 5 days). Thus, more than one patch may be required to provide continuous antiemetic prophylaxis. Characterisation of the pharmacokinetics of multiple transdermal dosing offers useful information for clinicians who treat patients with the latter types of regimens.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female Caucasian subjects
* Aged between 18 and 70 years, inclusive, at screening
* BMI between 20.0 and 29.9 kg/m², inclusive.
* Must demonstrate understanding of the purposes and risks of the study
* Must agree to follow the restrictions and schedule of study procedures

Exclusion Criteria:

* Current or previous disease, disorder, allergy or condition that could affect study conduct or laboratory assessments, or that presents undue risk from study medication or procedures.
* Physical examination or screening investigation result that indicates subject is unfit for the study.
* Scarring on upper arms.
* Positive virology, urine drugs of abuse or pregnancy test result (females of childbearing potential only).
* Recent use of prescribed or over the counter medication.
* Participation in any clinical study or loss of ≥ 400 mL of blood (e.g. been a blood donor) within the previous 60 days.
* Average weekly alcohol consumption of greater than 21 units (males) or 14 units (females), or habitually smokes ≥ 5 cigarettes or equivalent tobacco per day within the 6 months before the first study drug administration.
* Lactating female subjects and female subjects of childbearing potential who are not willing to use an acceptable form of contraception during and for 90 days after the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of the co-administration of IV granisetron and the Sancuso® patch | 0 to 336 hours post-dose

SECONDARY OUTCOMES:
Safety and tolerability of the coadministration of IV granisetron and the Sancuso® patch | Up to 28 days post-dose
Patch adhesion and residual granisetron after patch | 0 to 336 hours post-dose
Pharmacokinetic profile of repeated Sancuso® patch application | 0 to 336 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Mair, Principal Investigator — Syneos Health
Locations (1):
- Charles River Clinical Services Edinburgh Ltd, Edinburgh, United Kingdom